CLINICAL TRIAL: NCT02554318
Title: The Effect of Fermented Soybean Supplementation on the Body Weight and Physical Function of Tuberculosis Patients With Standard Therapy in Indonesia
Brief Title: Fermented Soybean Supplementation Among Active Pulmonary Tuberculosis Patients With Standard Therapy in Indonesia
Acronym: FSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Indonesian Directorate General of Higher Education (Other Government)
Responsible Party: Principal Investigator, Budhi Setiawan, dr, M.Kes, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DGHE 626/E4.4/K/2011
Record Dates: First submitted 2015-09-14; First posted 2015-09-18 (Estimated); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Tuberculosis; Body Weight Changes; Motor Activity
Keywords: Tempeh; Body weight; Handgrip strength; 6MWT; Supplementation; Wasting
MeSH Terms: conditions — Tuberculosis, Pulmonary; Body Weight Changes; Motor Activity; Body Weight; Cachexia | interventions — Rifampin; Isoniazid; Pyrazinamide; Ethambutol; Soy Foods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): TB standard therapy with fixed dose combination :
  once per day by mouth for 2 months Fixed dose combination = RHZE (150mg/75mg/400mg/275mg) R=rifampicin, H=isoniazid, Z=pyrazinamide, E=ethambutol,
  Patients with body weight: 30 - 37 kg = 2 tablets, 38 - 54 kg = 3 tablets, 55 - 70 kg = 4 tablets, and ≥71 kg = 5 tablets
  and 166.5 grams cooked fermented soybean (tempeh) daily for two months
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol; Dietary Supplement: Fermented soybean
- Control (Active Comparator): TB standard therapy with fixed dose combination :
  once per day by mouth for 2 months Fixed dose combination = RHZE (150mg/75mg/400mg/275mg) R=rifampicin, H=isoniazid, Z=pyrazinamide, E=ethambutol,
  Patients with body weight: 30 - 37 kg = 2 tablets, 38 - 54 kg = 3 tablets, 55 - 70 kg = 4 tablets, and ≥71 kg = 5 tablets
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol

INTERVENTIONS:
Drug: Rifampicin
  Other Names: Rifampin; Rifadin
Drug: Isoniazid
  Other Names: Hydra; Isovit
Drug: Pyrazinamide
  Other Names: Actizid; Cavizide
Drug: Ethambutol
  Other Names: Myambutol; Servambutol
Dietary Supplement: Fermented soybean
  Other Names: Tempeh
  Arms: Intervention

SUMMARY:
Tuberculosis (TB) patients often have a lower body mass index (BMI) and experience wasting. Wasting reduces lean body mass and may cause physical function impairment. This study aimed to determine the efficacy of fermented soybeans (tempeh) as a food supplement on body weight and physical function changes among active pulmonary tuberculosis patients with standard therapy.

DETAILED DESCRIPTION:
This study was carried out at the outpatient department building, lung hospital Surabaya, Indonesia. As a national health referral system in TB program, the hospital was related to four local sub district health centers that were involved in the recruitment of participants in the study.

Patients with newly diagnosed pulmonary tuberculosis were randomly assigned into two groups, namely intervention group, which consisted of 65 participants and control group which had 64 participants. Randomization was carried out using sealed, unmarked opaque envelopes that are allocated to participants in this study. A minimum sample size of per group (n=64) was determined by Windows version G*Power 3.1.5 software to identify a mean difference in body weight change of ≥1.1 kg between intervention and control groups.

The intervention group obtained the standard therapy of TB and an additional 166.5 grams of boiled tempeh daily for two months. The control group obtained only standard TB therapy. Patients in the intervention group were instructed to divide one cake tempeh into three pieces and eat them three times in a day. Consumption frequencies of supplements were recorded in a logbook by an enumerator during random visits once a week. One of the patient family members was asked to help to supervise compliance.

The participants were assessed before and after the intervention period for both groups. Body weight of the participants was evaluated by measuring the change in body weight. The change of physical function was assessed by handgrip strength using a digital dynamometer and 6-minute walk test (6MWT). Protein and caloric intakes were estimated twice, measured during the first and second months using 24-hour dietary recall method during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed adult male and female TB active patients
* Having clinical evidences of active TB symptoms
* Positive or negative sputum smears
* Having positive chest X-ray that compatible with a diagnosis of tuberculosis
* No history of previous anti tuberculosis treatment
* Give a written informed consent and basic contact data

Exclusion Criteria:

* Heavy smoker (> 20 cigarettes per day)
* Pregnancy and lactation
* Extra pulmonary TB
* Known allergy to soybean
* Having clinical evidences of any underlying disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Krawinkel, Prof. Dr., Study Director — University of Giessen

REFERENCES:
- [Background] Paton NI, Chua YK, Earnest A, Chee CB. Randomized controlled trial of nutritional supplementation in patients with newly diagnosed tuberculosis and wasting. Am J Clin Nutr. 2004 Aug;80(2):460-5. doi: 10.1093/ajcn/80.2.460. PMID 15277171
- [Background] Martins N, Morris P, Kelly PM. Food incentives to improve completion of tuberculosis treatment: randomised controlled trial in Dili, Timor-Leste. BMJ. 2009 Oct 26;339:b4248. doi: 10.1136/bmj.b4248. PMID 19858174
- [Background] Jahnavi G, Sudha CH. Randomised controlled trial of food supplements in patients with newly diagnosed tuberculosis and wasting. Singapore Med J. 2010 Dec;51(12):957-62. PMID 21221502
- [Background] PrayGod G, Range N, Faurholt-Jepsen D, Jeremiah K, Faurholt-Jepsen M, Aabye MG, Jensen L, Jensen AV, Grewal HM, Magnussen P, Changalucha J, Andersen AB, Friis H. The effect of energy-protein supplementation on weight, body composition and handgrip strength among pulmonary tuberculosis HIV-co-infected patients: randomised controlled trial in Mwanza, Tanzania. Br J Nutr. 2012 Jan;107(2):263-71. doi: 10.1017/S0007114511002832. Epub 2011 Jul 6. PMID 21729372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2013 and February 2015, patients who attended the lung clinics in Surabaya for newly diagnosed pulmonary TB were screened for study enrollment.
Pre-assignment Details: After the enrollment of the study, several participants withdrew their assignment due to several reasons such as underlying disease, heavy smoker, they did not stay in the city, plan to move to other city, and dislike the food.
Groups:
- Intervention: TB standard therapy with fixed dose combination :
  once per day by mouth for 2 months Fixed dose combination = RHZE (150mg/75mg/400mg/275mg) R=rifampicin, H=isoniazid, Z=pyrazinamide, E=ethambutol,
  Patients with body weight: 30 - 37 kg = 2 tablets, 38 - 54 kg = 3 tablets, 55 - 70 kg = 4 tablets, and ≥71 kg = 5 tablets
  and 166.5 grams cooked fermented soybean (tempeh) daily for two months
  Rifampicin
  Isoniazid
  Pyrazinamide
  Ethambutol
  Fermented soybean
- Control: TB standard therapy with fixed dose combination :
  once per day by mouth for 2 months Fixed dose combination = RHZE (150mg/75mg/400mg/275mg) R=rifampicin, H=isoniazid, Z=pyrazinamide, E=ethambutol,
  Patients with body weight: 30 - 37 kg = 2 tablets, 38 - 54 kg = 3 tablets, 55 - 70 kg = 4 tablets, and ≥71 kg = 5 tablets
  Rifampicin
  Isoniazid
  Pyrazinamide
  Ethambutol
Period: Overall Study
Arm/Group | Intervention | Control
Started | 75 | 72
Completed | 65 | 64
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 10 | 8

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population of the participants was assessed by age, gender, education, income, occupation, ethnicity, sputum smear examination result, and Body Mass Index.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 65 | 64 | 129
Age, Categorical [Count of Participants; unit: Participants] — Participants were newly diagnosed adult male and female pulmonary TB active patients aged between 18 and 55 years. Population: The number of Baseline Participants was assigned to the arm groups based on the inclusion and exclusion criteria. Some of them have rejected and withdrawn for some reasons such as objection and underlying diseases.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 65 | 64 | 129
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.11 (9.63) | 34.45 (10.35) | 32.77 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 35 | 35 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Javanese | 32 | 28 | 60
  Madurese | 31 | 34 | 65
  Others | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Indonesia: Surabaya, East Java | 65 | 64 | 129
  Indonesia: Others | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: Kg/m²] | 18.41 (3.10) | 18.57 (3.26) | 18.49 (3.17)
Education [Count of Participants; unit: Participants]
  Elementary School | 26 | 27 | 53
  Middle School | 12 | 8 | 20
  High school | 23 | 24 | 47
  Bachelor | 4 | 5 | 9
Income (million rupiahs) [Count of Participants; unit: Participants]
  Less than one | 38 | 37 | 75
  Between one to three | 26 | 27 | 53
  More than three | 1 | 0 | 1
Occupation [Count of Participants; unit: Participants]
  Unemployed | 19 | 22 | 41
  Part timer | 5 | 3 | 8
  Private | 41 | 39 | 80
Sputum Smear [Count of Participants; unit: Participants]
  Positive | 44 | 44 | 88
  Negative | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Bodyweight on a Digital Weight Scale From Baseline at 2 Months
Description: Change of body weight of the participants over the two months intervention period as measured on a kilograms scale. The change was calculated from two-time points as the value at the later time point minus the value at the earlier time point. Positive numbers represent increases and negative numbers represent decreases. A higher value score in change means a better outcome on nutritional status for the patients after the study.
Time Frame: Baseline, 2 months
Population: All participants were assessed their body weight (kg) using an electronic weight scale before and after the study to determine its change.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Intervention | Control
Number analyzed (Participants) | 65 | 64
Kilogram | 2.80 (2.33) | 1.44 (2.42)

2. Secondary Outcome: Change in Hand-grip Strength on a Digital Dynamometer Scale From Baseline at 2 Months
Description: The change of hand-grip strength of the participants over the two months intervention period was measured on a kilograms scale. The change was calculated from two-time points as the value at the later time point minus the value at the earlier time point. Positive numbers represent increases and negative numbers represent decreases. The higher scores reflected the better physical function outcomes of the patients.
Time Frame: Baseline, 2 months
Population: All participants were measured from two-times points, before and after the study in order to analyze their change after 2 months of intervention. Higher values reflected better physical function results.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | Intervention | Control
Number analyzed (Participants) | 65 | 64
Kilogram | 3.90 (4.50) | 0.84 (4.83)

3. Secondary Outcome: Change in Distance on 6-minute Walk Test (6MWT) From Baseline at 2 Months
Description: The change distance in meters scale as assessed by 6MWT according to American Thoracic Society (ATS) 2002 guidelines. The 6MWT was carried out on a track along the 30-meter corridor marked by two colored cones placed at both ends of the track alignment. The participants were asked using the standard instruction to walk at their self-selected pace back and forth between the cones as far as they could for 6 minutes. The distance taken by each participant was measured and then recorded. Instructions were given to every patient by reading a guideline with the same intonations to every patient before performing the test. The result of the 6MWT was expressed in meters. The change was calculated from two-time points as the value at the later time point minus the value at the earlier time point. Higher scores reflected better physical function outcomes.
Time Frame: Baseline, 2 months
Population: Not all participants were analyzed before and after the study to measure the change in the distance. Only 64 participants from the intervention group and 63 participants from the control group contributed to data collection.
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 64 | 63
Meter | 49.67 (58.49) | 25.75 (56.85)

4. Secondary Outcome: Change in Body Mass Index (BMI) From Baseline at 2 Months
Description: The change in BMI was assessed by a digital weight scale and height scale (kg/m²). The formula for BMI is weight in kilograms divided by height in meters squared. The change was calculated from two-time points as the value at the later time point minus the value at the earlier time point. Higher scores reflected the better nutritional status results of the patients.
Time Frame: Baseline, 2 months
Population: All participants were assessed before and after the study using a standard formula to determine the change of the body mass index (BMI).
Measure: Mean (Standard Deviation); unit: Kg/m²
Arm/Group | Intervention | Control
Number analyzed (Participants) | 65 | 64
Kg/m² | 1.13 (0.93) | 0.54 (0.94)

5. Other Pre Specified Outcome: Caloric Intake on 24-hour Dietary Recall Method at the 2nd and 6th.
Description: The average calorie intake (in kcal/day) was assessed by the 24-hour dietary recall questionnaire and calculated by NutriSurvey software version 2005, with the country-specific food database for Indonesia.
Time Frame: In the course of the 8 week intervention, two interviews were conducted; at the 2nd and 6th week.
Population: Not all participants were assessed their calorie intake, only 61 participants in the control arm and all participants from intervention contributed to the data collection.
Measure: Mean (Standard Deviation); unit: Kcal/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 65 | 61
Kcal/day
  2nd week | 1980.10 (437.79) | 1844.64 (592.13)
  6th week | 2227.98 (463.72) | 2059.27 (550.52)
  Average | 2113.16 (429.41) | 1972.12 (530.04)

6. Other Pre Specified Outcome: Protein Intake on 24-hour Dietary Recall Method.
Description: The average protein intake (in Gram/day) was assessed by the 24-hour dietary recall questionnaire and calculated using NutriSurvey software version 2005, with the country specific food database for Indonesia.
Time Frame: In the course of the 8 week intervention, two interviews were conducted; at the 2nd and 6th week.
Population: Not all participants were assessed before and after the study, only 61 participants from the control group contributed to the data collection of the study.
Measure: Mean (Standard Deviation); unit: Gram/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 65 | 61
Gram/day
  2nd week | 77.34 (27.98) | 69.49 (22.81)
  6th week | 77.70 (26.72) | 73.35 (24.37)
  Average | 77.52 (26.63) | 71.42 (21.06)

ADVERSE EVENTS:
Time Frame: The intervention period was 2 months for each participant who is eligible for the study. All participants were assessed at month zero (baseline) and month two (end line). The recruitment method was not a one-time event but a referral from physicians. Since eligible participants were not always available every day at the clinics thus the adverse data collection period for all participants was 1 year and 3 months.
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, are the same from the clinicaltrials.gov definitions. Observation for adverse event was done three times a week since the food should be delivered regularly and regular notes taken on a log book.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/72
Other Adverse Events (participants affected / at risk) | 1/75 | 0/72
OTHER ADVERSE EVENTS (reported when occurring in more than 0.013% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=75) | Control (N=72)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
It needs more participants and not all patients were tested for HIV since it was not suitable for the local culture. High temperature which is involved in the cooking process could change the chemical properties of tempeh. Since physical activity consists of complex aspects, a combination of several tools can be used in a study to give a comprehensive view of interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No